CLINICAL TRIAL: NCT07144735
Title: Allogeneic Gamma Delta (γδ) T Cells for the Treatment of Glioblastoma
Brief Title: Allogeneic γδT Cells in Glioblastoma
Acronym: ABOUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University (Other); Changping Laboratory (Other)
Responsible Party: Principal Investigator, Chenlong YANG, Research Professor, Peking University Third Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M20250397
Record Dates: First submitted 2025-08-14; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma (GBM); Glioblastoma Multiforme (GBM)
Keywords: Glioblastoma; Glioblastoma Multiforme; Immunotherapy; Gamma Delta T Cell; γδT
MeSH Terms: conditions — Glioblastoma | interventions — Cell Count

STUDY DESIGN:
Intervention Model Description: 3+3 Dose escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose (Experimental): Dose 1: 7x10^7 ABOUT γδT, local administration every 3-4 weeks
  Interventions: Drug: Allogeneic γδ T (ABOUT) cells
- Medium dose (Experimental): Dose 2: 1.1x10^8 ABOUT γδT, local administration every 3-4 weeks
  Interventions: Drug: Allogeneic γδ T (ABOUT) cells
- High dose (Experimental): Dose 3: 1.6x10^8 ABOUT γδT, local administration every 3-4 weeks
  Interventions: Drug: Allogeneic γδ T (ABOUT) cells

INTERVENTIONS:
Drug: Allogeneic γδ T (ABOUT) cells — Allogeneic γδ T cells genetically edited to knockout the ARIH1 and BCL11b genes.
  Other Names: ARIH1 and BCL11b knockout γδ T cells; ARIH1KO/BCL11bKO γδ T cells

SUMMARY:
This first-in-human clinical study aims to evaluate the safety and feasibility of locally delivered, allogeneic γδ T cells (genetically edited with ARIH1 and BCL11b knockout, designated ABOUT γδT cells) in patients with glioblastoma multiforme (GBM). The engineered effector cells are delivered via localized administration to selectively target and eliminate residual GBM cells. ABOUT: ARIH1 and BCL11b knockOUT γδ T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18-70 years old (both ends included)
2. At least one evaluable lesion with previous biopsy or pathohistologic confirmation of glioblastoma (WHO grade IV), with imaging suggestive of continued progression or recurrence after comprehensive treatment
3. Karnofsky Performance Status (KPS) ≥ 60%
4. Life expectancy > 4 weeks
5. Patients who completed radiotherapy or systemic therapies (including temozolomide/bevacizumab or other agents) for at least 4 weeks prior to enrollment. All prior treatment-related toxicities should be defined as ≤ grade 1 (except for toxicities such as alopecia or leukoplakia) according to the Common Terminology Standard for Adverse Events (CTCAE 6.0)
6. Must be able to undergo an MRI with contrast
7. Must have adequate organ and marrow function as defined below:

   * White blood cell count (WBC) ≥ 3 x 10^9/L
   * Absolute neutrophil count (ANC) > 1 x 10^9/L
   * Hemoglobin (Hb) ≥ 90 g/L
   * Platelet (PLT) ≥ 80×10^9/L
   * Albumin transaminase (ALT) & albumin transaminase (AST) < 1.5 × institutional upper limit of normal (ULN)
   * Serum creatinine (Cr) < 1.5 x institutional ULN
   * Total bilirubin < 1.5 x institutional ULN
   * PT & PTT ≤ 1.25 x institutional ULN
8. No obvious hereditary diseases
9. Normal cardiac function with left ventricular ejection fraction >55%
10. No bleeding and coagulation disorders
11. Absence of positive blood cultures for bacteria, fungus, or virus within 48-hours prior to ABOUT γδT cell infusion and/or there aren't any indications of meningitis
12. Fertile women must have had a pregnancy test with a negative result within 7 days prior to the start of treatment, and subjects are willing to use contraception (hormonal or barrier method of birth control or abstinence) during the clinical trial and for 6 months after the last cell infusion; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
13. Signed, written informed consent

Exclusion Criteria:

1. Active hepatitis B or C virus, HIV infection, or other untreated active infection
2. Pregnant and lactating women
3. Participants with organ failure
4. Participants with a chronic disease requiring immunologic or hormonal therapy
5. Participants with an allergy to immunotherapy and related cells
6. Participants with uncontrolled intercurrent illness
7. Participants with psychiatric illness/social situations that would limit compliance with study requirements
8. Participants with a history of organ transplantation or who are awaiting organ transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 3 months following ABOUT γδT cells administration
  Defined as the incidence of ≥ Grade 3-4 adverse events related to ABOUT γδT cells according to common terminology criteria for adverse events (CTCAE) v6.0.
Incidence of Dose-Limiting Toxicities (DLTs) | 28 days following initial treatment with ABOUT γδT cells
  Defined as events attributable to ABOUT γδT cells infusion within 28 days post-infusion. Grade 3-4 acute graft-versus-host disease (GvHD) according to the Mount Sinai Acute GvHD International Consortium criteria; Grade 3 or higher cytokine release syndrome (CRS) lasting more than 2 weeks, according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria; Any ABOUT γδT cells-related AE requiring intubation; Grade 4 non-hematologic toxicities.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 3 months following ABOUT γδT cells administration
  According to modified RANO criteria, ORR is defined as proportion of subjects with confirmed CR and PR.
Duration of response (DOR) | 3 months following ABOUT γδT cells administration
  According to modified RANO criteria, DOR is defined as time from the date when a response of confirmed CR/PR is first met to the date of confirmed disease progression or death.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhengzhou Second Hospital, Zhengzhou, Henan
  - Henan Academy of Innovations in Medical Science, Zhengzhou, Henan